CLINICAL TRIAL: NCT04135781
Title: Adjuvant Nab-paclitaxel Plus S-1 Versus Capecitabine Plus Oxaliplatin for Patients With Stage III Gastric Cancer After D2 Gastrectomy : a Randomised，Open-label, Phase III Study
Brief Title: Nab-paclitaxel Combined With S-1 as Adjuvant Chemotherapy for Stage Ⅲ Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xiangdong Cheng, Director, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-KAL-GC-04
Record Dates: First submitted 2019-10-20; First posted 2019-10-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Stomach Cancer
Keywords: nab-paclitaxel; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Taxes; Albumin-Bound Paclitaxel; Tegafur; S 1 (combination); Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AS (Experimental): Arm A：nab paclitaxel （120mg/m2；iv；d1，8）+S-1 （<1.25 m2, 40 mg; 1.25 to ≤1.5 m2, 50 mg; and ≥ 1.5 m2, 60 mg；po；d1-14 bid）Q3W；up to eight cycles
  Interventions: Drug: nab paclitaxel; Drug: Tegafur
- XELOX (Active Comparator): Arm B：Capetabine（1000 mg/m2 po, d1-14 bid ）+ Oxaliplatin（130mg/m2 , iv, d1）Q3W；up to eight cycles
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: nab paclitaxel — nab paclitaxel （120mg/m2；iv；d1，8）
  Other Names: albumin bound paclitaxel
  Arms: AS
Drug: Tegafur — S-1 （<1.25 m2, 40 mg; 1.25 to ≤1.5 m2, 50 mg; and ≥ 1.5 m2, 60 mg；po；d1-14 bid）
  Other Names: S-1
  Arms: AS
Drug: Oxaliplatin — Oxaliplatin（130mg/m2 , iv, d1）
  Arms: XELOX
Drug: Capecitabine — Capetabine（1000 mg/m2 po, d1-14 bid ）
  Arms: XELOX

SUMMARY:
This is a randomized, open-label phase III study. The treatment was compare the efficacy and safety of Albumin-bound Paclitaxel plus S-1 versus Oxaliplatin plus capecitabine (XELOX) treating stage Ⅲ gastric cancer as adjuvant setting

DETAILED DESCRIPTION:
This is a randomized, open-label phase III study. The treatment was compare the efficacy and safety of Albumin-bound Paclitaxel plus S-1 versus Oxaliplatin plus capecitabine (XELOX) treating stage Ⅲ gastric cancer as adjuvant setting. The primary endpoint is the 3-year diseases-free survival (DFS) rate. The secondary endpoints are the overall survival (OS) and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-75 years;
2. Histological diagnosis of stage III gastric adenocarcinoma and Gastroesophageal junction of the stomach;
3. Patients are required to provide a pathologically confirmed diagnosis report and provide 4-5 histological white films obtained at baseline;;
4. Patients underwent D2 radical resection within 6 weeks prior to random enrollment; and R0 resection criteria were achieved;
5. Ability to perform chemotherapy within 7 days of enrollment in the randomized group;
6. No prior anti-tumor treatment (including systemic chemotherapy and local radiotherapy), except for initial gastrectomy for primary lesions;
7. ECOG performance status of 0-1;
8. Haematological status: absolute neutrophil count(ANC) ≥1.5×109 /L, platelet count(PLT) ≥100×109 /L, hemoglobin(HB) ≥90 g/L;WBC ≥3.0×109 /L;And no bleeding tendency;
9. Liver function: alanine glutamate transaminase (ALT) and glutamate transaminase (AST) ≤2.5 x upper limit of normal range (ULN), alkaline phosphatase ≤2.5 x upper limit of normal range (ULN)；total bilirubin (TBIL)≤1.5 x upper limit of normal range (ULN), or≤3 x upper limit of normal range (ULN) when with Gilbert's syndrome;
10. kidney function: Creatinine(Cr)≤1.5 x upper limit of normal range(ULN) or Creatinine clearance >60 ml/min (calculated according to Cockroft-Gault)
11. Able and willing to comply with the study plans in this protocol and sign the informed consent;

Exclusion Criteria:

1. Treat with any other study drug or participate in another clinical trial with therapeutic intent within 28 days prior to enrollment;
2. postoperative complications requiring clinical intervention and affecting treatment, such as stomach cramps, dumping syndrome;
3. Patients known to be allergic or intolerant to clinical trial drugs;
4. investigator believes will affect the subject's treatment regimen, uncontrolled serious medical diseases, including severe heart disease (such as the New York Heart Association (NYHA) Level II or more Congestive heart failure), cerebrovascular disease, uncontrolled diabetes, uncontrolled high blood pressure, uncontrolled infection；
5. Known active infection with HIV, hepatitis B or hepatitis C;
6. Other serious and uncontrolled non-malignant disease; except adequately treated cervical carcinoma in situ, non-melanoma skin Localized prostate cancer after cancer and radical surgery (PSA ≤ 10 ng/ml); no recurrence or metastasis was found based on imaging follow-up results and any disease-specific tumor markers;
7. accompanied by dysphagia, complete or incomplete gastrointestinal obstruction, active gastrointestinal bleeding, perforation;
8. Female patients during pregnancy or lactation, who are refused to receive contraception during the childbearing age;
9. The investigator judges patients who are not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
3 years Diseases-free Survival rate(3 years-DFS) | up to 3 years
  DFS is defined as time from the date of inclusion up to the date of disease progression or death

SECONDARY OUTCOMES:
Overall survival (OS) | up to 3 years
  Overall survival is defined as time from the start of treatment until death due to any reason.
Safety as measured by number and grade of adverse events | up to 3 years
  Summary adverse events according to NCI-CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Cheng xiangdong, PhD, Study Chair — Zhejiang Cancer Hospital；Cancer hospital of the university of chinese academy of sciences
Locations (1):
- Zhejiang Cancer Hospital；Cancer hospital of the university of chinese academy of sciences, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng X, Wu D, Xu N, Chen L, Yan Z, Chen P, Zhou L, Yu J, Cui J, Li W, Wang C, Feng W, Wei Y, Yu P, Du Y, Ying J, Xu Z, Yang L, Zhang Y. Adjuvant albumin-bound paclitaxel combined with S-1 vs. oxaliplatin combined with capecitabine after D2 gastrectomy in patients with stage III gastric adenocarcinoma: a phase III multicenter, open-label, randomized controlled clinical trial protocol. BMC Cancer. 2021 Jan 12;21(1):56. doi: 10.1186/s12885-020-07772-7. PMID 33435909